CLINICAL TRIAL: NCT05242302
Title: Efficacy of End-to-Side Nerve Transfer for Patients With Severe Cubital Tunnel Syndrome
Brief Title: AIN Transfer for Cubital Tunnel Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00066610
Record Dates: First submitted 2022-01-31; First posted 2022-02-16 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2022-02

CONDITIONS: Nerve Injury; Surgery
Keywords: nerve transfer; cubital tunnel syndrome; nerve generation
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Nerve Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- reverse end to side nerve transfer (Experimental)
  Interventions: Procedure: nerve transfer
- end to end nerve transfer (Active Comparator)
  Interventions: Procedure: nerve transfer
- nerve decompression (Active Comparator)
  Interventions: Procedure: nerve transfer

INTERVENTIONS:
Procedure: nerve transfer — the anterior interosseous nerve will be used as a donor to reinnervation the injured ulnar nerve.

SUMMARY:
Ulnar nerve compressive injury due to cubital tunnel syndrome is very common. Because of the long distance to the target muscles in the hand, functional outcome in severe cases even with decompression surgery is often poor. Therefore, alternative treatment options are much needed. Recently, anterior interosseous nerve reverse end to side (RETS) transfer to the ulnar nerve above the wrist has gained popularity. However, whether a substantial portion of motor axons in the donor nerve are indeed capable of breaching the connective tissues in the ulnar nerve to reach the target muscles in the hand remains untested. To answer this crucial question, in this study the investigators plan to recruit 60 cubital tunnel syndrome patients with marked motor axonal loss who will undergo the RETS procedure. Motor unit number estimation will be done on the ulnar and anterior interosseous nerves at baseline and repeated at 3 and 6 months post operatively. Hand motor function and disability scores will also be tested at the same time points. Given the importance of this critical question and the potential utilities of distal nerve transfers, this should be a worthwhile effort.

DETAILED DESCRIPTION:
Introduction Peripheral nerve trauma especially through compressive injury is very common. Of these, ulnar neuropathy at the elbow is the second most prevalent. In severe cases, functional outcomes even with surgery are often poor. Principle reasons being that the ulnar nerve innervates a large number of intrinsic hand muscles. At an average of 350 mm from the site of injury to the target muscles, the distance is very long, Although peripheral nerve fibres have the ability to regenerate, it is very slow at only 1 mm/day. That would translate to a year for the regenerating fibres to reach the hand. With the favorable condition in the distal stump and target muscles to regrowth rapidly declining over time, few axons will successfully reach target. Therefore, alternative methods of surgical treatments are being sought to circumvent this major hurdle.

Rationale and purpose One potentially promising alternative is through distal nerve transfer by using a terminal branch of the anterior interosseous nerve (AIN) to the pronator quadratus muscle and coapt it to the ulnar nerve close to the wrist. That would greatly shorten the distance to target by 200 mm or more. By approximating the end of the AIN donor stump to the side of the ulnar nerve through an eipneurial window (termed reverse end to side or RETS) transfer, it allows preservation of the integrity of the ulnar nerve fibres thus providing a conduit for the regenerating native axons to reach the hand. While this concept is theoretically appealing and has gained increasing popularity in clinical practice, a crucial question of central importance remains answered: Can the AIN donor axons indeed breach the ulnar nerve trunk and reinnervate the hand muscles? Aside from testing the central premise of RETS, it would be important to know the exact magnitude of reinnervation that can be achieved from the donor nerve through this procedure.

With the above rationale in mind, the objective of this proposal is to test the hypothesis that reinnervation of ulnar intrinsic hand muscles by the AIN can be achieved through the RETS procedure. This will be done through quantifying the amount of innervation by the AIN donor nerve to the ulnar intrinsic hand muscles using motor unit number estimation, a non-invasive electrophysiological technique. The investigators will also evaluate whether there is an associated improvement in hand function following the procedure.

Experimental protocol Subjects For this study, the investigators aim to recruit a prospective series of 60 patients with severe cubital tunnel syndrome causing marked motor axonal loss.

Primary outcome measures Motor unit number estimations of native axons in the ulnar nerve innervation the intrinsic hand muscles compared to those from the AIN.

Secondary outcomes

Motor function:

i) Pinch strength using a pinch gauge ii) Grip strength using a Jamar dynamometer iii) Disabilities of Arm, Hand and Shoulder (DASH) Questionnaire

Procedures and follow up All outcomes will be measured at baseline and repeated at 3 and 6 months post op. Motor unit number estimation will be done using the multiple point stimulation technique. To briefly summarize, recording surface electrodes will be placed over the belly of the hypothenar muscles. To estimate the number of native ulnar axons innverating the hypothenar hand muscles, supramaximal stimulation of the ulnar nerve in the mid forearm above the site of AIN coaptation will be done. A sample of single motor unit action potentials will be obtained by discretely stimulating individual motor axons using finely graded stimuli. A motor unit number estimation will be calculated from the ratio of the compound muscle action potential amplitude and the average single motor unit action potentials. To estimate the motor unit innervation from the AIN, the same procedure will be done by stimulating the median nerve while recording from the hypothenar muscles.

Surgery Eligible patients will undergo surgical decompression of the ulnar nerve at the elbow. Additionally, a reverse end-to-side transfer to the ulnar nerve will be done using a terminal branch of the AIN to the pronator quadratus muscle. It will be coapted to the side of the motor fascicle of the ulnar nerve just above the wrist through a 5 mm epineurial window.

Statistical analysis To address the central question of AIN innervation, descriptive statistics (mean and sd) will be used to quantify the extent of nerve growth through the epineurial window created by the RETS procedure. Since there is no AIN innervation of the hypothenar muscles at baseline, growth of motor axons through the epineurial window should be easy to discern through motor unit number estimation. Changes in motor hand strength and disability following surgery will be compared using repaired measure one way ANOVA with time as the independent factor. With this being a pilot exploratory study, further analytic statistical analysis would not be justified as the sample size will be too small to allow for any meaningful interpretation.

Expected outcomes and significance This will be further aided by the very substantial distance difference between the entry point of the AIN to the ulnar nerve trunk at just above the wrist and the native ulnar motor axons that regenerate from the elbow. At less than 100 mm from the target muscles, many AIN motor axons should reach the hypothenar muscles by 3 months and all by 6 months. In contrast, the regenerating native ulnar motor axons would likely not reach the hand muscles for a year or more, as shown in the investigators' previous publications.

Given the importance of this critical question and the potential utilities of distal nerve transfers, this should be a worthwhile effort.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18)
* Symptoms and signs indicative of cubital tunnel syndrome
* Markedly depleted motor unit number estimate in the ulnar intrinsic hand muscles > 2 SD below the mean

Exclusion Criteria:

* Other co-existing neurological or musculoskeletal conditions affecting hand function
* Cognitive impairments rendering patient unable to follow instructions to perform functional tasks
* Unwilling to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Motor nerve conduction study | patients will be followed for 6 months after surgery
  Amplitudes of the maximum compound muscle action potentials evoked by median nerve stimulation

SECONDARY OUTCOMES:
Key pinch strength | patients will be followed for 6 months after surgery
  Dynamometer for isometric force quantification of pinch strength between the 1st and 2nd digits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No